CLINICAL TRIAL: NCT05227534
Title: A Prospective Multi-canceR Early-detection and interVENTional Study in Asymptomatic Individuals: PREVENT
Brief Title: Multi-canceR Early-detection Test in Asymptomatic Individuals (PREVENT)
Acronym: PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RSCD2022006
Record Dates: First submitted 2022-01-14; First posted 2022-02-07 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Cancer; Early Detection of Cancer; Circulating Cell-free DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants 40 years of age or older with cancer risk (Experimental): The study will aim to enroll participants 40 years of age or older with cancer risk. Specific cancer risks will be enriched to increase the number of cancer events that are observed during the study.
  Interventions: Device: OverC multi-cancer detection blood test

INTERVENTIONS:
Device: OverC multi-cancer detection blood test — Blood collection for the OverC multi-cancer detection blood test and standard-of-care screening with return of results

SUMMARY:
PREVENT is a prospective, multicenter, interventional study evaluating the performance of the OverC multi-cancer detection blood test in asymptomatic individuals with cancer risk.

DETAILED DESCRIPTION:
Participants will receive the OverC multi-cancer detection blood test along with standard-of-care screening, whose results will be returned to health care providers and participants. The diagnostic procedures will be guided firstly by the OverC multi-cancer detection blood test and then by the standard-of-care screening. The number, cancer types, and cancer clinical stage of cancer patients diagnosed via the OverC multi-cancer detection blood test will be recorded.

The study will enroll approximately 12,500 participants as defined by eligibility criteria with an anticipated enrollment period of approximately 9 months at up to 30 clinical sites within China. Participants will be actively followed for approximately 5 years from the date of their enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to provide a written informed consent form
* Participants must not have received any colonoscopy, abdominal MRI/CT, low-dose CT, or chest CT within 5 years before signing the informed consent form
* Participants must be able to provide blood samples for study tests
* Participants must be between 40 and 75 years old

Exclusion Criteria:

* Individuals who have an acute infection or inflammation within 14 days prior to recruitment
* Individuals with cancer-associated clinical symptoms or suspected of cancer
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
* Recipient of blood transfusion within 7 days prior to recruitment
* Individuals who have pure ground-glass opacity
* Unable to provide blood samples for the multi-cancer early detection blood test
* Individuals who are unable to tolerate standard-of-care cancer screening tests or have contraindications of standard-of-care cancer screening tests
* Individuals who have taken medication with anti-tumor effects within 30 days prior to recruitment
* Individuals who have received or are undergoing curative cancer treatment within three years prior to recruitment
* Individuals with hemorrhagic diseases
* Individuals with autoimmune diseases
* Individuals who are pregnant or lactating
* Individuals who have severe comorbidities that are not suitable for participating in the trial judged by researchers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The cancer clinical stages of cancer patients diagnosed via the multi-cancer detection blood test | Up to 5 years
Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) for the multi-cancer detection test alone or with standard-of-care screening as evaluated after 1-year follow-up | Up to 1 year

SECONDARY OUTCOMES:
Changes in health-related quality of life in individuals with a positive result of the multi-cancer detection test assessed by Short Form Health Survey (SF-12v2) | Up to 5 years
  The SF-12v2 is a measure of health related quality of life including physical component summary (PCS) and mental component summary (MCS). Both PCS and MCs have scores that range from 0 to 100. Higher values represent better health.
Changes in anxiety as evaluated by Self-rating Anxiety Scale (SAS) of individuals with a positive result of the multi-cancer detection test | Up to 5 years
  Assessed by Self-rating Anxiety Scale (SAS). Range in score from 25 to 100 with higher scores indicate greater severity of anxiety.
Satisfaction with the multi-cancer detection test | Up to 5 years
  Satisfaction will be measured by a self-reported questionnaire. Range in ranks from very satisfied, satisfied, general, unsatisfied, to very unsatisfied.
Sensitivity, specificity, PPV, and NPV for the multi-cancer detection blood test alone or with standard-of-care screening as evaluated after 3- and 5-year follow-up | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No